CLINICAL TRIAL: NCT06783855
Title: Outcomes of Uretheroileal Suspension Technique During Open Radical Cystectomy and Ileal Neobladder: A Prospective Randomized Comparative Study
Brief Title: Outcomes of Uretheroileal Suspension Technique During Open Radical Cystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdellah, assistant lecturer urology department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: soh-med-25-1-1MD
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Radical Cystectomy

STUDY DESIGN:
Intervention Model Description: This study will be conducted on 60 eligible patients The patients will be allocated into 2 groups: group (A) 30 patients will be treated with suspension uretheroileal technique and group (B) 30 patients will be treated without suspension technique act as control.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- : group (A) 30 patients will be treated with suspension uretheroileal technique (Active Comparator)
  Interventions: Procedure: suspension uretheroileal technique
- group (B) 30 patients will be treated with conventional radical cystectomy and ileal neobladder (Active Comparator)
  Interventions: Procedure: conventional radical cystectomy and ileal neobladder

INTERVENTIONS:
Procedure: suspension uretheroileal technique — The suspension technique is reported as the puboprostatic ligaments that attach the prostate to the symphysis pubis. After the ligating the complex, including both the dorsal vein complex and the puboprostatic ligaments, this complex was sharply divided anteriorly from the prostate with a safe distance (1-2 mm), and the urethra is defined and divided. After removing the prostate, the ileal pouch is reconstructed by completely everting the mucosa and sutured outward with a running 4-0 absorbable suture around the edge. The neck of the neobladder was narrowed to ≈1 cm, for convenient passage of a 20 F catheter. Anastomotic sutures of 3-0 absorbable polyglactin were placed at the 1, 3, 5, 6, 7, 9, 11 and 12 o'clock positions through the full thickness of the urethra
  Arms: : group (A) 30 patients will be treated with suspension uretheroileal technique
Procedure: conventional radical cystectomy and ileal neobladder — After removing the prostate, the ileal pouch is reconstructed by completely everting the mucosa and sutured outward with a running 4-0 absorbable suture around the edge. The neck of the neobladder was narrowed to ≈1 cm, for convenient passage of a 20 F catheter. Anastomotic sutures of 3-0 absorbable polyglactin were placed at the 1, 3, 5, 6, 7, 9, 11 and 12 o'clock positions through the full thickness of the urethra, including the mucosa and muscularis of the neobladder neck, ensuring mucosa-to-mucosa anastomosis
  Arms: group (B) 30 patients will be treated with conventional radical cystectomy and ileal neobladder

SUMMARY:
The suspension technique is reported as the puboprostatic ligaments that attach the prostate to the symphysis pubis. After the ligating the complex, including both the dorsal vein complex and the puboprostatic ligaments, this complex was sharply divided anteriorly from the prostate with a safe distance (1-2 mm), and the urethra is defined and divided. After removing the prostate, the ileal pouch is reconstructed by completely everting the mucosa and sutured outward with a running 4-0 absorbable suture around the edge. The neck of the neobladder was narrowed to ≈1 cm, for convenient passage of a 20 F catheter. Anastomotic sutures of 3-0 absorbable polyglactin were placed at the 1, 3, 5, 6, 7, 9, 11 and 12 o'clock positions

DETAILED DESCRIPTION:
The suspension technique is reported as the puboprostatic ligaments that attach the prostate to the symphysis pubis. After the ligating the complex, including both the dorsal vein complex and the puboprostatic ligaments, this complex was sharply divided anteriorly from the prostate with a safe distance (1-2 mm), and the urethra is defined and divided. After removing the prostate, the ileal pouch is reconstructed by completely everting the mucosa and sutured outward with a running 4-0 absorbable suture around the edge. The neck of the neobladder was narrowed to ≈1 cm, for convenient passage of a 20 F catheter. Anastomotic sutures of 3-0 absorbable polyglactin were placed at the 1, 3, 5, 6, 7, 9, 11 and 12 o'clock positions through the full thickness of the urethra, including the mucosa and muscularis of the neobladder neck, ensuring mucosa-to-mucosa anastomosis. The sutures at the 1 and 11 o'clock positions were anchored to the ligated complex including both the dorsal vein complex and the puboprostatic ligaments, to suspend the poucho-urethral anastomosis (suspension technique). The difference between the suspension and no-suspension techniques is only the placing of two sutures into the ligated complex

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 years.
* Muscle-invasive bladder carcinoma (MIBC).
* Non-muscle-invasive bladder carcinoma (NMIBC) fulfilling the following criteria:

  1. - (recurrent disease that is unresponsive to other treatments
  2. - high-grade tumors (T1, carcinoma in situ) refractory to intravesical therapy
  3. -Multifocal or recurrent high-grade tumors despite intravesical therapy and the tumor progression from NMIBC to MIBC).

Exclusion Criteria:

* NMIBC or benign disease.
* Severe hepatic renal dysfunction.
* Urethral involvement with bladder carcinoma.
* Poor overall health status.
* Severe renal dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The continence rates at 1, 3, 6 and 12 months after the procedure will be evaluated | at 1, 3, 6 and 12 months after the procedure will be evaluated
  Urinary continence after urethroileal suspension technique

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt